CLINICAL TRIAL: NCT04097288
Title: Effects of Single Dose Citalopram and Reboxetine on Urethral and Anal Closure Function on Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Thea Christoffersen, Investigator, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSRI-UPR-01; 2019-000059-14 (EudraCT Number)
Record Dates: First submitted 2019-05-21; First posted 2019-09-20 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Stress Urinary Incontinence; Fecal Incontinence
Keywords: stress urinary incontinence; pharmacologic treatment; fecal incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Fecal Incontinence | interventions — Citalopram; Reboxetine

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, placebo controlled, three period cross over phase I study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Single dose citalopram (Experimental): A blinded single dose 40 mg citalopram is administered three hours before urethral pressure reflectometry and anal acoustic reflectometry measurements
  Interventions: Drug: Citalopram 40mg
- Single dose reboxetine (Active Comparator): A blinded single dose 8 mg reboxetine is administered two hours before urethral pressure reflectometry and anal acoustic reflectometry measurements
  Interventions: Drug: Reboxetine 8 mg
- Single dose placebo citalopram (Placebo Comparator): A blinded single dose visually identical placebo pill to citalopram is administered three hours before urethral pressure reflectometry and anal acoustic reflectometry measurements
  Interventions: Drug: Placebo oral tablet
- Single dose placebo reboxetine (Placebo Comparator): A blinded single dose visually identical placebo pill to reboxetine is administered two hours before urethral pressure reflectometry and anal acoustic reflectometry measurements
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Citalopram 40mg — Single dose
  Arms: Single dose citalopram
Drug: Reboxetine 8 mg — Single dose
  Arms: Single dose reboxetine
Drug: Placebo oral tablet — Single dose
  Other Names: Placebo to citalopram
  Arms: Single dose placebo citalopram
Drug: Placebo oral tablet — Single dose
  Other Names: Placebo tó reboxetine
  Arms: Single dose placebo reboxetine

SUMMARY:
This study will investigate if citalopram, a selective serotonin reuptake inhibitor, is reducing the opening pressure of the urethra and possibly causing or worsening stress urinary incontinence. Reboxetine, a norepinephrine reuptake inhibitor, is known to increase urethral opening pressure through actions on adrenoceptors in Onuf´s nucleus and will act as an active control.

Furthermore, this study is performed to explore the effects of reboxetine and citalopram on the opening pressure of the anal canal.

DETAILED DESCRIPTION:
This study will investigate if citalopram, a selective serotonin reuptake inhibitor, is reducing the opening pressure of the urethra and possibly causing or worsening stress urinary incontinence. Theoretically, citalopram can affect the tone of urethra through actions on serotonergic receptors in Onuf´s nucleus that innervates the striated muscle in urethra. Treatment with selective serotonin reuptake inhibitors is common and has been associated with urinary incontinence. Stress urinary incontinence is frequent and the most common cause of urinary incontinence. Reboxetine, a norepinephrine reuptake inhibitor, is known to increase urethral opening pressure through actions on adrenoceptors in Onuf´s nucleus and will act as an active control. Should the tone of urethra decrease significantly after ingestion of citalopram, this study would contribute to a deeper understanding of stress urinary incontinence and give rise to a debate of pharmacologic treatment of stress urinary incontinence diagnosed in patients treated with citalopram (this debate may also include use of selective serotonin reuptake inhibitor).

Furthermore, this study is performed to explore the effects of reboxetine and citalopram on the opening pressure of the anal canal. Onuf´s nucleus, like the striated urethral sphincter, innervates the striated skeletal muscle of the external sphincter in the anal canal. The prevalence of fecal incontinence (FI) increases with age and is estimated to affect 15% of people aged over 50 years. Pharmacologic treatment of fecal incontinence is very sparse and new treatments it is very desirable. If reboxetine or citalopram increases the anal opening pressure these pharmacologic agents might leads to new ways of treating FI, making this study the first to explore this area.

The design is a single center, randomized, double-blind, placebo controlled, three period cross over phase I study. Twenty-four healthy, female subjects are recruited and investigated during three independent trial days where one of the pharmacologic agents is given each trial day (citalopram, reboxetine or placebo) in concordance with the sequence (order of the pharmacologic agents given). Subjects will be drafted randomly and evenly among the three sequences possible. During all trial days pressures of the urethra and the anal canal of every subject will be measured by urethral pressure reflectometry and anal acoustic reflectometry at the time of maximum plasma concentration of citalopram and reboxetine. A clinically meaningful difference in urethral pressure after administration of citalopram is assessed to be 10 cmH2O compared to placebo (reboxetine acts as an active control) while a clinically meaningful difference in anal pressure after administration of citalopram or reboxetine is assessed to be 15 cmH2O compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent of participation
* Female
* Age between 18 and 55 years (both included)
* Normal weight (BMI 18,5 to 30,0 kg/m2).
* Regular use of safe contraceptive products ie. Intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long acting injections) through the entire trial and until eight days after the study has ended for the subject (registered at trial day one, two and three). Subjects who are postmenopausal (defined as no menses for 12 months or more prior enrolment) can be included without use of contraceptive products.

Exclusion Criteria:

* Known hypersensitivity of Citalopram.
* Known hypersensitivity of Edronax.
* A history of significant cardiovascular, gastrointestinal, endocrine, hematologic, immunologic, metabolic or genitourologic disease (including pelvic surgery because of trauma, pelvic trauma, lower urinary tract surgery, irradiation to the pelvis, history or evidence of an anatomical anomaly of the lower urinary tract, urinary outlet obstruction, urinary retention, urethral hypermobility , prolapse of pelvic organs, hematuria or urinary tract infection at screening) or lung disease, neurologic, dermatologic, psychiatric disease, kidney disease, malign diseases or other major diseases assessed by the investigator.
* Known QT-interval prolongation or congenital long QT syndrome
* History or objective symptoms of urinary incontinence
* Current infectious disease (fever and symptoms associated with viral or bacterial disease (including respiratory tract infections) or fungal disease (excluding cutaneous infection).
* Pulse under 40 beats pr. minute or above 100 beats pr. minute. Average systolic blood pressure above 140 mmHg or average diastolic blood pressure over 90 mmHg (average of three measurements performed on screening). In case blood pressure or pulse should deviate from these criteria allowance of three additional measurements are accepted.
* Current participation in other clinical trials that might affect the results of this trial (judged by the investigators).
* Use of prescription drugs, over the-counter drugs or herbalism drugs. Exceptions from these criteria are use of paracetamol (4 g a day) and safe contraception as stated above.
* Current consumption of alcohol above 14 units of alcohol a week.
* Smoking within three months.
* Drug abuse within three months.
* Present pregnancy, at screening or during the trial, including a positive pregnancy test (presented at trial day one, two or three).
* Breastfeeding at screening or during the study (registered at trial day one, two and three).
* Any kind of condition (anamnestic or objective) that the investigator assess that must lead to exclusion of this study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Difference in average UOP-placebo and average UOP-citalopram (during relaxation) | UPR measurements are performed 3 hours after blinded administration of citalopram or placebo to citalopram and two hours after blinded administration of reboxetine/placebo to reboxetine
  Difference in urethral opening pressure
Difference in average AOP-placebo and average AOP-citalopram or average AOP-reboxetine (during relaxation) | UPR measurements are performed 3 hours after blinded administration of citalopram or placebo to citalopram and two hours after blinded administration of reboxetine/placebo to reboxetine
  Difference in urethral opening pressure

SECONDARY OUTCOMES:
Difference in average UOP-placebo and average UOP-reboxetine (during relaxation) | UPR measurements are performed 3 hours after blinded administration of citalopram or placebo to citalopram and two hours after blinded administration of reboxetine/placebo to reboxetine
  Difference in urethral opening pressure
Difference in average UOP-placebo and average UOP-citalopram or UOP-reboxetine (during voluntary contraction) | UPR measurements are performed 3 hours after blinded administration of citalopram or placebo to citalopram and two hours after blinded administration of reboxetine/placebo to reboxetine
  Difference in urethral opening pressure
Difference in average AOP-placebo and average AOP-citalopram or AOP-reboxetine (during voluntary contraction). | UPR measurements are performed 3 hours after blinded administration of citalopram or placebo to citalopram and two hours after blinded administration of reboxetine/placebo to reboxetine
  Difference in urethral opening pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Sonne, DMSc, Principal Investigator — University Hospital Frederiksberg and Bispebjerg
Locations (1):
- Department of Clinical Pharmacology, Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No